CLINICAL TRIAL: NCT03445559
Title: A Multi-modal, Physician-centered Intervention to Improve Guideline-concordant Prostate Cancer Imaging
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 15-356; HX002038 (Other Grant/Funding Number: VA HSR&D)
Record Dates: First submitted 2018-02-20; First posted 2018-02-26 (Actual); Results first posted 2025-02-14 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Imaging; Veterans Affairs; Guideline Adherence; Implementation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: The proposed behavioral intervention will be implemented according to a stepped wedge cluster-randomized design. This is a single direction cross-over randomized trial where every site serves, at some point, as both a control and an intervention site. The first time point will be a baseline measurement, where none of the study sites have yet received the intervention. At subsequent time points, study sites initiate the intervention. The time at which each site initiates implementation of the intervention is randomized.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): No intervention
- Intervention (Experimental): The intervention is comprised of three components: 1) Clinical Order Check, 2) Academic Detailing, and 3) Audit and Feedback.
  Interventions: Behavioral: Clinical Order Check; Behavioral: Academic Detailing; Behavioral: Audit and Feedback

INTERVENTIONS:
Behavioral: Clinical Order Check — A Clinical Order Check is an evidence-based, systems-level method to affect significant behavior change. It addresses the intervention functions of education, enablement and incentivization which are effective methods to change behaviors driven by beliefs about capabilities, knowledge, social influences, beliefs about consequences, and environmental context and resources. All VA facilities currently use locally adapted clinical reminders. This strategy is technologically simple, straightforward, and is considered to be a best practice within the VA IT community. The reminder will be self-explanatory and non-intrusive to workflow.
  Arms: Intervention
Behavioral: Academic Detailing — Academic detailing is an individual and facility-level intervention consistently shown to improve provider behavior. This strategy addresses the intervention functions of persuasion, coercion, modeling, and education which are effective methods for affecting behaviors driven by beliefs about capabilities, knowledge, social influences, beliefs about consequences, and environmental context and resources. During the meeting, the detailer will follow a script explaining that the visit is part of an experimental program to provide physicians with up-to-date, unbiased information about imaging to stage prostate cancer.
  Arms: Intervention
Behavioral: Audit and Feedback — Audit and feedback is an effective, individual-level intervention for changing healthcare provider behavior, resulting in small but potentially clinically important benefits. Audit and feedback addresses the intervention functions of education, persuasion and incentivization, all of which are important for addressing beliefs about capabilities and consequences, knowledge, and social influence.
  Arms: Intervention

SUMMARY:
The primary aim of this study is to determine whether a multi-modal, physician-focused behavioral intervention can improve facility-level guideline-concordant utilization of prostate cancer staging imaging. Other aims of this study include to use mixed methods to explore physician influence on guideline-concordant imaging and to determine the cost and cost impact of a physician-focused behavioral intervention to improve guideline-concordant prostate cancer imaging.

DETAILED DESCRIPTION:
Almost half of Veterans with localized prostate cancer (the most common non-cutaneous malignancy among US men) receive inappropriate, wasteful imaging. The VHA Blueprint for Excellence prioritizes increasing operational effectiveness. Prior studies seeking to limit inappropriate imaging did not assess barriers and achieved mixed results. The investigators' team has explored the causes of guideline-discordant prostate cancer imaging and found that 1) patients with newly diagnosed prostate cancer have little concern for radiographic staging but rather focus on treatment, 2) physician trust imaging guidelines but are apt to follow their own intuition, fear medico-legal consequences, and succumb to influence from colleagues who image frequently. In spite of such discrepant views, most VHA physicians suggested or supported a large-scale effort to improve imaging use across VHA.

The investigators propose a multi-site, stepped wedge, cluster-randomized trial to determine the effect of a physician-focused behavioral intervention on VHA prostate cancer imaging use. The multi-level intervention, developed according to the Theoretical Determinants Framework, combines traditional physician behavior change methods with novel methods of communication and data collection. The intervention consists of three components: 1) a system of audit and feedback to clinicians informing individual clinicians and their sites about how their behavior compares to their peers' and to published guidelines 2) a program of academic detailing with the goal to educate providers about prostate cancer imaging, and 3) a CPRS Clinical Order Check for potentially inappropriate imaging. The intervention will be introduced to 10 participating geographically-distributed study sites.

The investigators will assess imaging rates 6 months prior to the intervention and 3 months following the intervention. The study's specific aims seek to understand the effects of the intervention on 1) facility-level prostate cancer imaging rates, 2) physician experience with and perceptions of the intervention and its implementation, and 3) the costs of both implementing the intervention and affecting change in imaging use. These aims will support a subsequent intervention to improve guideline-concordant imaging across VHA. Experience gained through this project will be leveraged to improve guideline-concordant care and increase operational effectiveness in other domains.

ELIGIBILITY:
Inclusion Criteria:

Provider Criteria:

* Urology Chiefs and attending urologists employed through the VA (full time, part time) at one of the 10 participating sites
* Physician Assistants and Nurse Practitioners employed through the VA at one of the 10 participating sites that work in the respective urology clinics
* Providers may be any gender or race/ethnicity

Qualitative portion only:

* Urology Chiefs and/or frontline staff physicians
* participating PAs & NPs having cared for at least 5 men with incident prostate cancer within the previous 6 months
* Patients will not be directly recruited into the study.
* The investigators have obtained a waiver of HIPAA authorization and informed consent to analyze electronic health records of patients that are diagnosed with ICD-9 code 185 or ICD-10 code C61 during the study period at the 10 participating sites.

Exclusion Criteria:

Provider Criteria:

* Urology Residents will be excluded.

Patients

* Patients will be excluded if they have a history of prior malignancy
* Are over the age of 85
* Diagnosed at autopsy or by death certificate
* Died within 3 months of diagnosis
* Not having data on at least one of the following:

  * PSA
  * clinical stage
  * Gleason score

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2026-02-28 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Danil V Makarov, MD MHS, Principal Investigator — VA NY Harbor Healthcare System, New York, NY
Locations (11):
- United States (11):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - VA NY Harbor Healthcare System, New York, NY, New York, New York
  - Syracuse VA Medical Center, Syracuse, NY, Syracuse, New York
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington
  - William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Makarov DV, Holmes-Rovner M, Rovner DR, Averch T, Barry MJ, Chrouser K, Gee WF, Goodrich K, Haynes M, Krahn M, Saigal C, Sox HC, Stacey D, Tessier C, Waterhouse RL, Fagerlin A. Quality Improvement Summit 2016: Shared Decision Making and Prostate Cancer Screening. Urol Pract. 2018 Nov;5(6):444-451. doi: 10.1016/j.urpr.2017.11.005. Epub 2017 Dec 4. PMID 37312342
- [Background] Skokan AJ, Dobbs RW, Harris AM, Tessier CD, Sajadi KP, Talwar R, Berger I, Guzzo TJ, Ziemba JB. Implementing a patient safety culture survey to identify and target process improvements in academic ambulatory urology practices: a multi-institutional collaborative. Can J Urol. 2020 Feb;27(1):10087-10092. PMID 32065864
- [Background] Ziemba JB, Tessier CD, Harris AM. Patient safety education and perceptions of safety culture in American and Canadian urological residency training programs. Can J Urol. 2020 Dec;27(6):10431-10436. PMID 33325343
- [Background] Hsiang W, Han X, Jemal A, Nguyen KA, Shuch B, Park H, Yu JB, Gross CP, Davidoff AJ, Leapman MS. The Association Between the Affordable Care Act and Insurance Status, Stage and Treatment in Patients with Testicular Cancer. Urol Pract. 2020 Jul;7(4):252-258. doi: 10.1097/upj.0000000000000109. Epub 2020 Jul 1. PMID 34017908
- [Background] Grinberg AS, Sellinger JJ, Sprenkle PC, Bandin AJ, Nawaf CB, Syed JS, Leapman MS. Effect of Diaphragmatic Breathing on Procedural Anxiety During Transrectal Prostate Biopsy. Urology. 2020 Mar;137:26-32. doi: 10.1016/j.urology.2019.12.024. Epub 2019 Dec 29. PMID 31893532
- [Background] Abello A, Leapman M, Kenney PA. Chasing the Pack: Association between Urology Hospital Rankings and Surgical Outcome. J Urol. 2020 May;203(5):890-891. doi: 10.1097/JU.0000000000000710. Epub 2019 Dec 20. No abstract available. PMID 32068499
- [Background] You H, Shang W, Min X, Weinreb J, Li Q, Leapman M, Wang L, Tian J. Sight and switch off: Nerve density visualization for interventions targeting nerves in prostate cancer. Sci Adv. 2020 Feb 5;6(6):eaax6040. doi: 10.1126/sciadv.aax6040. eCollection 2020 Feb. PMID 32076639
- [Background] Rajwa P, Hopen P, Mu L, Paradysz A, Wojnarowicz J, Gross CP, Leapman MS. Online Crowdfunding Response to Coronavirus Disease 2019. J Gen Intern Med. 2020 Aug;35(8):2482-2484. doi: 10.1007/s11606-020-05896-x. Epub 2020 May 27. No abstract available. PMID 32462566
- [Background] Ghabili K, Park HS, Yu JB, Sprenkle PC, Kim SP, Nguyen KA, Ma X, Gross CP, Leapman MS. National trends in the management of patients with positive surgical margins at radical prostatectomy. World J Urol. 2021 Apr;39(4):1141-1151. doi: 10.1007/s00345-020-03298-6. Epub 2020 Jun 19. PMID 32562045
- [Background] Leapman MS, Presley CJ, Zhu W, Soulos PR, Adelson KB, Miksad RA, Boffa DJ, Gross CP. Association of Programmed Cell Death Ligand 1 Expression Status With Receipt of Immune Checkpoint Inhibitors in Patients With Advanced Non-Small Cell Lung Cancer. JAMA Netw Open. 2020 Jun 1;3(6):e207205. doi: 10.1001/jamanetworkopen.2020.7205. PMID 32511721
- [Background] Hsiang WR, Honig S, Leapman MS. Evaluation of Online Telehealth Platforms for Treatment of Erectile Dysfunction. J Urol. 2021 Feb;205(2):330-332. doi: 10.1097/JU.0000000000001378. Epub 2020 Sep 18. No abstract available. PMID 32945730
- [Background] Salazar MC, Canavan ME, Walters SL, Herrin J, Schwartz JL, Leapman M, Boffa DJ. Evaluation of Cancer Care After Medicaid Expansion Under the Affordable Care Act. JAMA Netw Open. 2020 Sep 1;3(9):e2017544. doi: 10.1001/jamanetworkopen.2020.17544. PMID 32990734
- [Background] Miccio JA, Talcott WJ, Jairam V, Park HS, Yu JB, Leapman MS, Johnson SB, King MT, Nguyen PL, Kann BH. Quantifying treatment selection bias effect on survival in comparative effectiveness research: findings from low-risk prostate cancer patients. Prostate Cancer Prostatic Dis. 2021 Jun;24(2):414-422. doi: 10.1038/s41391-020-00291-3. Epub 2020 Sep 28. PMID 32989262
- [Background] Becker DJ, Rude T, Walter D, Wang C, Loeb S, Li H, Ciprut S, Kelly M, Zeliadt SB, Fagerlin A, Lepor H, Sherman S, Ravenell JE, Makarov DV. The Association of Veterans' PSA Screening Rates With Changes in USPSTF Recommendations. J Natl Cancer Inst. 2021 May 4;113(5):626-631. doi: 10.1093/jnci/djaa120. PMID 32797212
- [Background] Lane GI, Ellimoottil C, Wallner L, Lenherr S, Clemens JQ. Patient Reported Shared Decision Making in Urology from the Surgical Consumer Assessment of Healthcare Providers and Systems (CAHPS) Survey. Urol Pract. 2021 May;8(3):341-347. doi: 10.1097/UPJ.0000000000000216. Epub 2020 Dec 28. PMID 37145663
- [Result] Kirk PS, Borza T, Caram MEV, Shumway DA, Makarov DV, Burns JA, Shelton JB, Leppert JT, Chapman C, Chang M, Hollenbeck BK, Skolarus TA. Characterising potential bone scan overuse amongst men treated with radical prostatectomy. BJU Int. 2019 Jul;124(1):55-61. doi: 10.1111/bju.14551. Epub 2018 Nov 12. PMID 30246937
- [Result] Ciprut SE, Kelly MD, Walter D, Hoffman R, Becker DJ, Loeb S, Sedlander E, Tenner CT, Sherman SE, Zeliadt SB, Makarov DV. A Clinical Reminder Order Check Intervention to Improve Guideline-concordant Imaging Practices for Men With Prostate Cancer: A Pilot Study. Urology. 2020 Nov;145:113-119. doi: 10.1016/j.urology.2020.05.101. Epub 2020 Jul 25. PMID 32721517
- [Result] Makarov DV, Ciprut S, Kelly M, Walter D, Shedlin MG, Braithwaite RS, Tenner CT, Gold HT, Zeliadt S, Sherman SE. Protocol: A multi-modal, physician-centered intervention to improve guideline-concordant prostate cancer imaging. Trials. 2021 Oct 18;22(1):711. doi: 10.1186/s13063-021-05645-3. PMID 34663435
- [Derived] Makarov DV, Thomas JK, Ciprut S, Rivera AJ, Sherman SE, Braithwaite RS, Best SL, Blakely S, D'Agostino LA, Dahm P, Dash A, Leapman MS, Leppert JT, Sanchez A, Shelton JB, Tessier CD, Tenner CT, Gold HT, Shedlin MG, Zeliadt SB. Prostate Cancer Imaging Stewardship: a multimodal, physician-centered intervention for guideline-concordant imaging. J Natl Cancer Inst. 2025 Nov 1;117(11):2308-2316. doi: 10.1093/jnci/djaf210. PMID 40796156

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates: March 2018 - March 2021 Type of location: VA Medical Centers Urology providers (physicians, physician assistants, nurse practitioners) from 10 VA medical centers who treat prostate cancer were enrolled in the study. Prostate cancer patient charts were reviewed but were not directly recruited into the study.
Pre-assignment Details: There was a minimum 3 month (maximum 30 month) run-in period prior to provider exposure to the intervention. A total of 58 clinical providers were enrolled at 10 VAMC sites.
  At the 10 VAMC sites, 2,374 patient charts were reviewed, 2,358 met inclusion criteria and were assigned to an arm. 16 patient charts were excluded at baseline due to
  * Prior diagnosis of prostate cancer
  * History of other prior malignancy
  * Low risk & missing clinical stage or PSA
Groups:
- Sequence Site 1: 3 Months of Control, Then 33 Months of Intervention; Sequence Site 2: 6 Months of Control, Then 30 Months of Intervention; Sequence Site 3: 9 Months of Control, Then 27 Months of Intervention; Sequence Site 4: 12 Months of Control, Then 24 Months of Intervention; Sequence Site 5: 15 Months of Control, Then 21 Months of Intervention; Sequence Site 6: 18 Months of Control, Then 18 Months of Intervention; Sequence Site 7: 21 Months of Control, Then 15 Months of Intervention; Sequence Site 8: 24 Months of Control, Then 12 Months of Intervention; Sequence Site 9: 27 Months of Control, Then 9 Months of Intervention; Sequence Site 10: 30 Months of Control, Then 6 Months of Intervention: Control: No intervention. Patient charts reviewed prior to intervention initiation in stepped wedge design.
  Intervention: Patient charts reviewed after intervention initiation for guideline-concordant prostate cancer imaging. The intervention is comprised of three components: 1) Clinical Order Check, 2) Academic Detailing, and 3) Audit and Feedback.
Period: Step 0: Mar 2018 to May 2018
Arm/Group | Sequence Site 1: 3 Months of Control, Then 33 Months of Intervention | Sequence Site 2: 6 Months of Control, Then 30 Months of Intervention | Sequence Site 3: 9 Months of Control, Then 27 Months of Intervention | Sequence Site 4: 12 Months of Control, Then 24 Months of Intervention | Sequence Site 5: 15 Months of Control, Then 21 Months of Intervention | Sequence Site 6: 18 Months of Control, Then 18 Months of Intervention | Sequence Site 7: 21 Months of Control, Then 15 Months of Intervention | Sequence Site 8: 24 Months of Control, Then 12 Months of Intervention | Sequence Site 9: 27 Months of Control, Then 9 Months of Intervention | Sequence Site 10: 30 Months of Control, Then 6 Months of Intervention
Started (By pretrial design, all sites in Control during step 0 through May 2018, and step 1 began on June 2018 with first site randomized to intervention.) | 30 | 25 | 10 | 30 | 17 | 41 | 24 | 9 | 27 | 8
Completed | 30 | 25 | 10 | 30 | 17 | 41 | 24 | 9 | 27 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Step 1: June 2018 to Aug 2018
Arm/Group | Sequence Site 1: 3 Months of Control, Then 33 Months of Intervention | Sequence Site 2: 6 Months of Control, Then 30 Months of Intervention | Sequence Site 3: 9 Months of Control, Then 27 Months of Intervention | Sequence Site 4: 12 Months of Control, Then 24 Months of Intervention | Sequence Site 5: 15 Months of Control, Then 21 Months of Intervention | Sequence Site 6: 18 Months of Control, Then 18 Months of Intervention | Sequence Site 7: 21 Months of Control, Then 15 Months of Intervention | Sequence Site 8: 24 Months of Control, Then 12 Months of Intervention | Sequence Site 9: 27 Months of Control, Then 9 Months of Intervention | Sequence Site 10: 30 Months of Control, Then 6 Months of Intervention
Started | 33 | 33 | 23 | 27 | 23 | 38 | 20 | 11 | 25 | 17
Completed | 33 | 33 | 23 | 27 | 23 | 38 | 20 | 11 | 25 | 17
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Step 2: Sept 2018 to Nov 2018
Arm/Group | Sequence Site 1: 3 Months of Control, Then 33 Months of Intervention | Sequence Site 2: 6 Months of Control, Then 30 Months of Intervention | Sequence Site 3: 9 Months of Control, Then 27 Months of Intervention | Sequence Site 4: 12 Months of Control, Then 24 Months of Intervention | Sequence Site 5: 15 Months of Control, Then 21 Months of Intervention | Sequence Site 6: 18 Months of Control, Then 18 Months of Intervention | Sequence Site 7: 21 Months of Control, Then 15 Months of Intervention | Sequence Site 8: 24 Months of Control, Then 12 Months of Intervention | Sequence Site 9: 27 Months of Control, Then 9 Months of Intervention | Sequence Site 10: 30 Months of Control, Then 6 Months of Intervention
Started | 11 | 38 | 4 | 25 | 14 | 39 | 15 | 6 | 31 | 16
Completed | 11 | 38 | 4 | 25 | 14 | 39 | 15 | 6 | 31 | 16
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Step 3: Dec 2018 to Feb 2019
Arm/Group | Sequence Site 1: 3 Months of Control, Then 33 Months of Intervention | Sequence Site 2: 6 Months of Control, Then 30 Months of Intervention | Sequence Site 3: 9 Months of Control, Then 27 Months of Intervention | Sequence Site 4: 12 Months of Control, Then 24 Months of Intervention | Sequence Site 5: 15 Months of Control, Then 21 Months of Intervention | Sequence Site 6: 18 Months of Control, Then 18 Months of Intervention | Sequence Site 7: 21 Months of Control, Then 15 Months of Intervention | Sequence Site 8: 24 Months of Control, Then 12 Months of Intervention | Sequence Site 9: 27 Months of Control, Then 9 Months of Intervention | Sequence Site 10: 30 Months of Control, Then 6 Months of Intervention
Started | 28 | 23 | 19 | 28 | 14 | 26 | 19 | 10 | 22 | 20
Completed | 28 | 23 | 19 | 28 | 14 | 26 | 19 | 10 | 22 | 20
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Step 4: Mar 2019 to May 2019
Arm/Group | Sequence Site 1: 3 Months of Control, Then 33 Months of Intervention | Sequence Site 2: 6 Months of Control, Then 30 Months of Intervention | Sequence Site 3: 9 Months of Control, Then 27 Months of Intervention | Sequence Site 4: 12 Months of Control, Then 24 Months of Intervention | Sequence Site 5: 15 Months of Control, Then 21 Months of Intervention | Sequence Site 6: 18 Months of Control, Then 18 Months of Intervention | Sequence Site 7: 21 Months of Control, Then 15 Months of Intervention | Sequence Site 8: 24 Months of Control, Then 12 Months of Intervention | Sequence Site 9: 27 Months of Control, Then 9 Months of Intervention | Sequence Site 10: 30 Months of Control, Then 6 Months of Intervention
Started | 24 | 51 | 15 | 41 | 21 | 37 | 13 | 12 | 28 | 29
Completed | 24 | 51 | 15 | 41 | 21 | 37 | 13 | 12 | 28 | 29
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Step 5: June 2019 to Aug 2019
Arm/Group | Sequence Site 1: 3 Months of Control, Then 33 Months of Intervention | Sequence Site 2: 6 Months of Control, Then 30 Months of Intervention | Sequence Site 3: 9 Months of Control, Then 27 Months of Intervention | Sequence Site 4: 12 Months of Control, Then 24 Months of Intervention | Sequence Site 5: 15 Months of Control, Then 21 Months of Intervention | Sequence Site 6: 18 Months of Control, Then 18 Months of Intervention | Sequence Site 7: 21 Months of Control, Then 15 Months of Intervention | Sequence Site 8: 24 Months of Control, Then 12 Months of Intervention | Sequence Site 9: 27 Months of Control, Then 9 Months of Intervention | Sequence Site 10: 30 Months of Control, Then 6 Months of Intervention
Started | 23 | 22 | 9 | 31 | 25 | 34 | 18 | 8 | 22 | 14
Completed | 23 | 22 | 9 | 31 | 25 | 34 | 18 | 8 | 22 | 14
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Step 6: Sept 2019 to Nov 2019
Arm/Group | Sequence Site 1: 3 Months of Control, Then 33 Months of Intervention | Sequence Site 2: 6 Months of Control, Then 30 Months of Intervention | Sequence Site 3: 9 Months of Control, Then 27 Months of Intervention | Sequence Site 4: 12 Months of Control, Then 24 Months of Intervention | Sequence Site 5: 15 Months of Control, Then 21 Months of Intervention | Sequence Site 6: 18 Months of Control, Then 18 Months of Intervention | Sequence Site 7: 21 Months of Control, Then 15 Months of Intervention | Sequence Site 8: 24 Months of Control, Then 12 Months of Intervention | Sequence Site 9: 27 Months of Control, Then 9 Months of Intervention | Sequence Site 10: 30 Months of Control, Then 6 Months of Intervention
Started | 27 | 33 | 13 | 29 | 17 | 34 | 21 | 8 | 20 | 13
Completed | 27 | 33 | 13 | 29 | 17 | 34 | 21 | 8 | 20 | 13
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Step 7: Dec 2019 to Feb 2020
Arm/Group | Sequence Site 1: 3 Months of Control, Then 33 Months of Intervention | Sequence Site 2: 6 Months of Control, Then 30 Months of Intervention | Sequence Site 3: 9 Months of Control, Then 27 Months of Intervention | Sequence Site 4: 12 Months of Control, Then 24 Months of Intervention | Sequence Site 5: 15 Months of Control, Then 21 Months of Intervention | Sequence Site 6: 18 Months of Control, Then 18 Months of Intervention | Sequence Site 7: 21 Months of Control, Then 15 Months of Intervention | Sequence Site 8: 24 Months of Control, Then 12 Months of Intervention | Sequence Site 9: 27 Months of Control, Then 9 Months of Intervention | Sequence Site 10: 30 Months of Control, Then 6 Months of Intervention
Started | 17 | 26 | 5 | 35 | 10 | 39 | 14 | 9 | 24 | 24
Completed | 17 | 26 | 5 | 35 | 10 | 39 | 14 | 9 | 24 | 24
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Step 8: Mar 2020 to May 2020
Arm/Group | Sequence Site 1: 3 Months of Control, Then 33 Months of Intervention | Sequence Site 2: 6 Months of Control, Then 30 Months of Intervention | Sequence Site 3: 9 Months of Control, Then 27 Months of Intervention | Sequence Site 4: 12 Months of Control, Then 24 Months of Intervention | Sequence Site 5: 15 Months of Control, Then 21 Months of Intervention | Sequence Site 6: 18 Months of Control, Then 18 Months of Intervention | Sequence Site 7: 21 Months of Control, Then 15 Months of Intervention | Sequence Site 8: 24 Months of Control, Then 12 Months of Intervention | Sequence Site 9: 27 Months of Control, Then 9 Months of Intervention | Sequence Site 10: 30 Months of Control, Then 6 Months of Intervention
Started | 6 | 19 | 3 | 11 | 9 | 9 | 6 | 11 | 18 | 5
Completed | 6 | 19 | 3 | 11 | 9 | 9 | 6 | 11 | 18 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Step 9: June 2020 to Aug 2020
Arm/Group | Sequence Site 1: 3 Months of Control, Then 33 Months of Intervention | Sequence Site 2: 6 Months of Control, Then 30 Months of Intervention | Sequence Site 3: 9 Months of Control, Then 27 Months of Intervention | Sequence Site 4: 12 Months of Control, Then 24 Months of Intervention | Sequence Site 5: 15 Months of Control, Then 21 Months of Intervention | Sequence Site 6: 18 Months of Control, Then 18 Months of Intervention | Sequence Site 7: 21 Months of Control, Then 15 Months of Intervention | Sequence Site 8: 24 Months of Control, Then 12 Months of Intervention | Sequence Site 9: 27 Months of Control, Then 9 Months of Intervention | Sequence Site 10: 30 Months of Control, Then 6 Months of Intervention
Started | 11 | 8 | 8 | 22 | 8 | 8 | 13 | 12 | 22 | 10
Completed | 11 | 8 | 8 | 22 | 8 | 8 | 13 | 12 | 22 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Step 10: Sept 2020 to Nov 2020
Arm/Group | Sequence Site 1: 3 Months of Control, Then 33 Months of Intervention | Sequence Site 2: 6 Months of Control, Then 30 Months of Intervention | Sequence Site 3: 9 Months of Control, Then 27 Months of Intervention | Sequence Site 4: 12 Months of Control, Then 24 Months of Intervention | Sequence Site 5: 15 Months of Control, Then 21 Months of Intervention | Sequence Site 6: 18 Months of Control, Then 18 Months of Intervention | Sequence Site 7: 21 Months of Control, Then 15 Months of Intervention | Sequence Site 8: 24 Months of Control, Then 12 Months of Intervention | Sequence Site 9: 27 Months of Control, Then 9 Months of Intervention | Sequence Site 10: 30 Months of Control, Then 6 Months of Intervention
Started | 23 | 23 | 24 | 27 | 8 | 22 | 19 | 11 | 8 | 25
Completed | 23 | 23 | 24 | 27 | 8 | 22 | 19 | 11 | 8 | 25
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Step 11: Dec 2020 to Feb 2021
Arm/Group | Sequence Site 1: 3 Months of Control, Then 33 Months of Intervention | Sequence Site 2: 6 Months of Control, Then 30 Months of Intervention | Sequence Site 3: 9 Months of Control, Then 27 Months of Intervention | Sequence Site 4: 12 Months of Control, Then 24 Months of Intervention | Sequence Site 5: 15 Months of Control, Then 21 Months of Intervention | Sequence Site 6: 18 Months of Control, Then 18 Months of Intervention | Sequence Site 7: 21 Months of Control, Then 15 Months of Intervention | Sequence Site 8: 24 Months of Control, Then 12 Months of Intervention | Sequence Site 9: 27 Months of Control, Then 9 Months of Intervention | Sequence Site 10: 30 Months of Control, Then 6 Months of Intervention
Started (By pretrial design: Step 11: 3 months of Intervention) | 20 | 22 | 17 | 27 | 11 | 25 | 21 | 15 | 10 | 9
Completed | 20 | 22 | 17 | 27 | 11 | 25 | 21 | 15 | 10 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control - Bone Scan Imaging Not Indicated: Patient charts reviewed prior to intervention initiation in a stepped wedge design where a bone scan was not indicated according to National Comprehensive Cancer Network guidelines.
- Intervention - Bone Scan Imaging Not Indicated: Patient charts reviewed after intervention initiation where a bone scan was not indicated according to National Comprehensive Cancer Network guidelines.
  The intervention is comprised of three components: 1) Clinical Order Check, 2) Academic Detailing, and 3) Audit and Feedback.
  Clinical Order Check: A Clinical Order Check is an evidence-based, systems-level method to affect significant behavior change. It addresses the intervention functions of education, enablement and incentivization which are effective methods to change behaviors driven by beliefs about capabilities, knowledge, social influences, beliefs about consequences, and environmental context and resources.
  Academic Detailing: Academic detailing is an individual and facility-level intervention consistently shown to improve provider behavior. This strategy addresses the intervention functions of persuasion, coercion, modeling, and education which are effective methods for affecting behaviors driven by beliefs about capabilities, knowledge, social influences, beliefs about consequences, and environmental context and resources.
  Audit and Feedback: Audit and feedback is an effective, individual-level intervention for changing healthcare provider behavior. Audit and feedback addresses the intervention functions of education, persuasion and incentivization, all of which are important for addressing beliefs about capabilities and consequences, knowledge, and social influence.
- Control - Bone Scan Imaging Indicated: Patient charts reviewed prior to intervention initiation in a stepped wedge design where a bone scan was indicated according to National Comprehensive Cancer Network guidelines.
- Intervention - Bone Scan Imaging Indicated: Patient charts reviewed after intervention initiation where a bone scan was indicated according to National Comprehensive Cancer Network guidelines.
- Intervention - Providers: Enrolled Urology Providers (urologists, Physician Assistants, Nurse Practitioners) who treat prostate cancer patients at the 10 participating VA Medical Centers.
  The following baseline characteristics were not collected from enrolled providers: 1) Reside in Zip Code with High Education, 2) Reside in Zip Code with High Broadband Access, and 3) Marital Status.
- Total: Total of all reporting groups
Arm/Group | Control - Bone Scan Imaging Not Indicated | Intervention - Bone Scan Imaging Not Indicated | Control - Bone Scan Imaging Indicated | Intervention - Bone Scan Imaging Indicated | Intervention - Providers | Total
Number analyzed (Participants) | 690 | 734 | 425 | 453 | 58 | 2360
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.9 (12.6) | 66.7 (6.8) | 68.0 (10.3) | 67.2 (10.5) | 49.71 (5.09) | 67.3 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data for measure was not entered by 4 providers in survey.
  Participants
    number analyzed (Participants) | 690 | 734 | 425 | 453 | 54 | 2356
    Female | 0 | 0 | 0 | 0 | 10 | 10
    Male | 690 | 734 | 425 | 453 | 44 | 2346
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Black | 531 | 538 | 329 | 301 | 55 | 1754
  Black | 116 | 138 | 56 | 84 | 3 | 397
  Not reported | 43 | 58 | 40 | 68 | 0 | 209
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 690 | 734 | 425 | 453 | 58 | 2360
Reside in Zip Code with High Education [Count of Participants; unit: Participants] — A Zip Code population with more than 20% of civilians with a Bachelor's degree or higher was classified as a high education zip code. Population: Data measure not collected for enrolled providers.
  Participants
    number analyzed (Participants) | 690 | 734 | 425 | 453 | 0 | 2302
    (all) | 485 | 524 | 306 | 280 |  | 1595
Reside in Zip Code with High Broadband Access [Count of Participants; unit: Participants] — Population: Data measure not collected for enrolled providers.
  Participants
    number analyzed (Participants) | 690 | 734 | 425 | 453 | 0 | 2302
    (all) | 616 | 604 | 368 | 350 |  | 1938
Marital Status [Count of Participants; unit: Participants] — Population: Data measure not collected for enrolled providers.
  Participants
    Not currently married: number analyzed (Participants) | 690 | 734 | 425 | 453 | 0 | 2302
    Not currently married | 307 | 361 | 215 | 216 |  | 1099
    Married: number analyzed (Participants) | 690 | 734 | 425 | 453 | 0 | 2302
    Married | 372 | 345 | 198 | 189 |  | 1104
    Not reported: number analyzed (Participants) | 690 | 734 | 425 | 453 | 0 | 2302
    Not reported | 11 | 28 | 12 | 48 |  | 99

OUTCOME MEASURES:

1. Primary Outcome: Facility-level Inappropriate Prostate Cancer Bone Scan Imaging Rates
Description: Facility-level utilization of bone scan imaging among men with newly diagnosed, low-risk prostate cancer. (Inappropriate Imaging according to NCCN guidelines)
Time Frame: Through study completion, an average of 4 years
Measure: Count of Participants; unit: Participants
Groups:
- Control: No intervention. Patient charts reviewed prior to intervention initiation in stepped wedge design.
- Intervention: Patient charts reviewed after intervention initiation for guideline-concordant prostate cancer imaging.
  The intervention is comprised of three components: 1) Clinical Order Check, 2) Academic Detailing, and 3) Audit and Feedback.
  Clinical Order Check: A Clinical Order Check is an evidence-based, systems-level method to affect significant behavior change. It addresses the intervention functions of education, enablement and incentivization which are effective methods to change behaviors driven by beliefs about capabilities, knowledge, social influences, beliefs about consequences, and environmental context and resources.
  Academic Detailing: Academic detailing is an individual and facility-level intervention consistently shown to improve provider behavior. This strategy addresses the intervention functions of persuasion, coercion, modeling, and education which are effective methods for affecting behaviors driven by beliefs about capabilities, knowledge, social influences, beliefs about consequences, and environmental context and resources.
  Audit and Feedback: Audit and feedback is an effective, individual-level intervention for changing healthcare provider behavior. Audit and feedback addresses the intervention functions of education, persuasion and incentivization, all of which are important for addressing beliefs about capabilities and consequences, knowledge, and social influence.
Arm/Group | Control | Intervention
Number analyzed (Participants) | 690 | 734
Participants | 141 | 109
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = 0.006, Chi-squared; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.30 to 0.98]

2. Primary Outcome: Facility-level Appropriate Prostate Cancer Bone Scan Imaging Rates
Description: Facility-level utilization of bone scan imaging among men with newly diagnosed, high-risk prostate cancer. (Appropriate Imaging according to NCCN guidelines)
Time Frame: Through study completion, an average of 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 425 | 453
Participants | 396 | 428
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = 0.42, Chi-squared; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.70 to 2.66]

3. Secondary Outcome: Individual-level Inappropriate Prostate Cancer Imaging Rates
Description: Provider-level utilization of nuclear medicine bone scan among men with newly diagnosed, low-risk prostate cancer (Inappropriate Imaging). Imaging is not recommended to stage low-risk prostate cancer men with PSA<10, Gleason<7, and clinical stage <T3.
Time Frame: Through study completion, an average of 4 years
Population: Clinical provider encounters (urologists, nurse practitioners, and physician assistants) that can order imaging for staging of prostate cancer patients. Patients may have seen multiple unique providers during the study period.
Measure: Median (Inter-Quartile Range); unit: percentage of inappropriate bone scans
Arm/Group | Control | Intervention
Number analyzed (Participants) | 77 | 68
percentage of inappropriate bone scans | 10.7 [8 to 19] | 8 [0 to 14]
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; Median Difference (Final Values) = 2.7

4. Secondary Outcome: Individual-level Appropriate Prostate Cancer Imaging Rates
Description: Provider-level utilization of bone scan or abdominal/pelvic CT or abdominal/pelvic MRI among men with newly diagnosed, high-risk prostate cancer. (Appropriate Imaging)
Time Frame: Through study completion, an average of 4 years
Reporting Status: Not Posted, anticipated posting 2026-02

5. Secondary Outcome: Provider Attitudes Regarding Prostate Cancer Imaging Guidelines and the Behavioral Intervention
Description: Qualitative outcome assessed through semi-structured, in-depth interviews with participating providers
Time Frame: Through study completion, an average of 4 years
Reporting Status: Not Posted, anticipated posting 2026-02

ADVERSE EVENTS:
Time Frame: Adverse event data were monitored for 6 months post-enrollment for all participants throughout the study.
Groups:
- Intervention Providers: Enrolled Urology Providers (urologists, Physician Assistants, Nurse Practitioners) who treat prostate cancer patients at the 10 participating VA Medical Centers.
Arm/Group | Control | Intervention | Intervention Providers
All-Cause Mortality (participants affected / at risk) | 1/1149 | 1/1267 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/1149 | 0/1267 | 0/58
Other Adverse Events (participants affected / at risk) | 0/1149 | 0/1267 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/59/NCT03445559/Prot_SAP_000.pdf